CLINICAL TRIAL: NCT00710931
Title: Visual Function With Bilateral AcrySof® ReSTOR® Aspheric SN6AD1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCONsur001.08
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Cataract
Keywords: Bilateral Cataract; IOL; ReSTOR; Aspheric
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReSTOR +3 Multifocal Lens (Experimental): Bilateral implantation of the AcrySof ReSTOR +3 Intraocular Lens (IOL)
  Interventions: Device: AcrySof ReSTOR Aspheric IOL model SN6AD1

INTERVENTIONS:
Device: AcrySof ReSTOR Aspheric IOL model SN6AD1 — Bilateral implantation of the AcrySof ReSTOR +3 Intraocular Lens (IOL) following cataract removal.

SUMMARY:
The objective of this study is to prospectively evaluate the visual parameters in a series of patients after phacoemulsification cataract surgery in a series of patients bilaterally implanted with the AcrySof® ReSTOR® Aspheric +3.0 Intraocular Lens (IOL).

ELIGIBILITY:
Inclusion Criteria:

* Prospective subjects should be 21 years of age and older, be of any race and gender and meet study entry criteria. Subject must require extraction of cataracts followed by implantation of a posterior chamber intraocular lens (IOL). Subjects must be candidates for bilateral removal of the natural crystalline lens followed by implantation of a multifocal IOL and be willing and able to complete all follow-up visits.

Exclusion Criteria:

* Subjects with pre-existing conditions that could skew the results or are contraindications for the AcrySof® ReSTOR® IOL should be excluded from the study. Please consult the AcrySof® ReSTOR® Aspheric product inserts under "Precautions" for subject groups that should be excluded from this study.

All subjects must have ≤ 0.75 diopters of astigmatism preoperatively as measured by Keratometry (K) readings. If the surgeon determines that a correction of cylinder is necessary postoperatively, this may be performed after the three month evaluations are completed.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ReSTOR +3 Multifocal Lens
Started | 34
Completed | 29
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | ReSTOR +3 Multifocal Lens
Number analyzed (Participants) | 34
Age Continuous [Median (Standard Deviation); unit: years] | 74.5 (6.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Binocular Visual Acuity at Distance, Near and Intermediate
Description: Uncorrected and best corrected visual acuity (VA) was tested at 4 meters (m), 60 centimeters (cm), and near at preferred distance (distance chosen by each subject and recorded in cm; mean and standard deviation calculated) with a standard ETDRS chart for distance and a hand held chart for near. VA is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better VA.
Time Frame: 6 months after surgery
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | ReSTOR +3 Multifocal Lens
Number analyzed (Participants) | 34
LogMAR
  Uncorrected VA at 4 m | 0.00 (0.08)
  Uncorrected VA at 60 cm | 0.13 (0.11)
  Uncorrected VA best near (39.69 cm +/- 4.09 cm) | 0.07 (0.08)
  Best Corrected VA at 4 m | 0.00 (0.06)
  Best Corrected VA at 60 cm | 0.09 (0.11)
  Best Corrected VA best near (41.31 cm +/- 5.82 cm) | 0.07 (0.08)

ADVERSE EVENTS:
Description: Adverse events were not collected in this study.
Arm/Group | ReSTOR +3 Multifocal Lens
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
When a clinical study report or manuscript, in lieu of a final report, is completed, Alcon will provide the summary findings of the study to the investigator.